CLINICAL TRIAL: NCT04234828
Title: Validation of the Diagnostic Performance of the Withings Sleep Device in Detecting Sleep Apnea Syndrome
Brief Title: Validation of Withings Sleep for the Detection of Sleep Apnea Syndrome
Acronym: VPASS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A00977-50
Record Dates: First submitted 2019-12-11; First posted 2020-01-21 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-01

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep Apnea; Sleep Apnea Syndromes; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory; Signs and Symptoms; Sleep Apnea, Obstructive; Sleep Disorders, Intrinsic; Dyssomnias; Sleep Wake Disorders; Nervous System Diseases; Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory; Signs and Symptoms; Sleep Apnea, Obstructive; Sleep Disorders, Intrinsic; Dyssomnias; Sleep Wake Disorders; Nervous System Diseases; Apnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred for an overnight in-lab PSG: Simultaneous assessment of SAS with Withings Sleep Device and overnight PSG

SUMMARY:
Sleep Apnea Syndrome (SAS) is a common pathology affecting between 4 and 8% of the general population. It aggravates morbidity and cardio-metabolic mortality and is responsible for accidents related to vigilance disorders. It is estimated that 80% of SAS cases are not diagnosed and therefore not treated. It is however impracticable to propose a diagnostic test of polygraphy (PG) or polysomnography (PSG) to every patient because of the cost and insufficient availability of these exams. It would therefore be useful to carry out a screening test before directing the patient to a complete test.

Several simplified polygraph systems with 2 or 3 channels have been proposed (nasal cannula, oximetry, heart rate) but they generally record only one night and remain intrusive enough to perturb the sleep.

The Withings Sleep is a non-contact device, along with an airbag placed under the mattress, which allows screening of SAS from four signals: movement, breathing, heart rate and snoring. The objective of the present study is to validate the diagnostic performance of the Withings Sleep for the detection of SAS compared to PSG.

ELIGIBILITY:
Inclusion Criteria:

* adults, men or women, aged between 18 and 70
* patients referred for an overnight polysomnographic exam for a suspicion of sleep-disordered breathing

Exclusion Criteria:

* children less than 18 years of age
* patients treated with continuous positive airway pressure
* person not giving her consent
* vulnerable subject according to current regulation:
* pregnant woman, parturient or breastfeeding
* subject deprived of freedom by judicial, medical or administrative decision
* subject legally protected or unable to express his consent
* subject non-beneficiary of healthcare
* subject falling into more than one of the above categories
* subject in linguistic or psychic incapacity to express his consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for an in-lab PSG exam
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of Withings Sleep at AHI threshold value of 15/h in PSG | immediately after intervention
  Sensitivity and specificity for SAS detection by Withings Sleep compared to polysomnography (PSG) at apnea-hypopnea index (AHI) threshold value of 15/h in PSG.
Sensitivity and specificity of Withings Sleep at AHI threshold value of 30/h in PSG | immediately after intervention
  Sensitivity and specificity for SAS detection by Withings Sleep compared to PSG at AHI threshold value of 30/h in PSG.

SECONDARY OUTCOMES:
Sensitivity and specificity of polygraphy (PG) | immediately after intervention
  Sensitivity and specificity for SAS detection by polygraphy (PG) compared to PSG at AHI threshold values of 15/h in PSG.
Sensitivity and specificity of PG | immediately after intervention
  Sensitivity and specificity for SAS detection by PG compared to PSG at AHI threshold values of 30/h in PSG.
Accuracy of Withings Sleep to estimate total sleep time (TST) given by PSG | immediately after intervention
  Bias and mean absolute error (MAE)
Accuracy of Withings Sleep to estimate sleep efficiency (SE) given by PSG | immediately after intervention
  Bias and MAE
Accuracy of Withings Sleep to estimate wake after sleep onset (WASO) given by PSG | immediately after intervention
  Bias and MAE
Influence of the position of the sleeper (decubitus dorsal vs decubitus latero-ventral) on the error of the AHI predicted by Withings Sleep compared with PSG | immediately after intervention
  Mean group difference between sleepers more than 50% of TST in decubitus dorsal or not.
Impact of the proportion of hypopnea events on the performance of Withings Sleep | immediately after intervention
  Mean group difference between patients with a majority of apnea events and patients with a majority of hypopnea events.
Mean group difference between patients with central or mixed apnea and patients with obstructive apnea events. | immediately after intervention
  Mean group difference between patients with a majority of central or mixed apnea events and patients with a majority of obstructive apnea events.
Reliability of Withings Sleep | immediately after intervention
  Rate of unusable or lost nights.
Reliability of PSG | immediately after intervention
  Rate of unusable or lost nights.

CONTACTS AND LOCATIONS:
Overall Officials: Garbiel Roisman, Principal Investigator — Hôpital Antoine Béclère
Locations (2):
- Service de pneumologie - Laboratoire du sommeil - CHU St-Pierre, Brussels, Belgium
- Service Explorations Fonctionnelles - Centre de Médecine du Sommeil - Hôpital Antoine Béclère, Clamart, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edouard P, Campo D, Bartet P, Yang RY, Bruyneel M, Roisman G, Escourrou P. Validation of the Withings Sleep Analyzer, an under-the-mattress device for the detection of moderate-severe sleep apnea syndrome. J Clin Sleep Med. 2021 Jun 1;17(6):1217-1227. doi: 10.5664/jcsm.9168. PMID 33590821